CLINICAL TRIAL: NCT07173478
Title: A Multicenter, Randomized, Double-blind, Vehicle-controlled, Parallel-group Comparison Trial to Demonstrate the Superiority of 1% OPA-15406 Foam to the Vehicle in Adult Patients With Atopic Dermatitis (Phase 3 Trial)
Brief Title: A Phase 3 Trial to Demonstrate the Superiority of 1% OPA-15406 Foam to the Vehicle in Adult Patients With Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 271-102-00043
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — difamilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1% OPA-15406 foam (Experimental)
  Interventions: Drug: OPA-15406
- Vehicle (Experimental)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OPA-15406 — 1% foam, topical, twice daily, for 4 weeks
  Other Names: difamilast
  Arms: 1% OPA-15406 foam
Drug: Vehicle — vehicle, topical, twice daily, for 4 weeks
  Arms: Vehicle

SUMMARY:
To investigate the superiority of 1% OPA-15406 foam to the vehicle in adult patients with atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been diagnosed AD based on the Diagnostic Criteria for Atopic Dermatitis (Criteria of the Japanese Dermatological Association)
* Participants with a history of AD for at least 3 years
* Participants who have an affected area covering from 5% to 40% of their body surface area (excluding the scalp) at the screening and baseline examinations
* Participants with an IGA score of 2 or 3 at the screening and baseline examinations

Exclusion Criteria:

* Participants who experienced an acute exacerbation of AD or contact dermatitis within 28 days prior to the baseline examination
* Participants who have been treated with OPA-15406 ointment in the past

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Success rate in Investigator's Global Assessment (IGA) | Week 4
  The investigator or subinvestigator assessed the skin symptoms using IGA. The investigator or subinvestigator scored the severity (0 = clear, 1 = almost clear, 2 =mild, 3 = moderate, 4 = severe/very severe) of the overall symptoms of the treatment area (erythema, infiltration, papules, effusion and scab formation) from baseline to Week 4. Incidence of success in IGA is defined as the rate of participants whose IGA score is 0 (clear) or 1 (almost clear) and has improved by at least 2 grades (responders) from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhito Sanada, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Mita Dermatology Clinic, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.